CLINICAL TRIAL: NCT04049747
Title: Imperial Prostate 4: Comparative Health Research Outcomes of NOvel Surgery in Prostate Cancer
Brief Title: Comparative Health Research Outcomes of NOvel Surgery in Prostate Cancer
Acronym: IP4-CHRONOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Prostate Cancer UK (Other); Imperial Clinical Trials Unit (ICTU) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19CX5006
Record Dates: First submitted 2019-06-04; First posted 2019-08-08 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Non-metastatic Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate Cancer; prostate adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Prostatectomy; Brachytherapy; Cryotherapy; WW Domain-Containing Oxidoreductase; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Two linked Randomised Controlled Trials with CHRONOS-A and CHRONOS-B discussed with patients and choice of A or B dependent on physician and patient equipoise.
  * CHRONOS-A Two arm RCT
  * CHRONOS-B Multi-Arm Multi-Stage (MAMS) Randomised Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- CHRONOS A - Arm 1 (Control) (Experimental): Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy]). In patients undergoing radiotherapy a maximum of 6-months neo-adjuvant hormonal therapy will be allowed. In patients undergoing radical prostatectomy, cytoreduction of maximum 6 months with medication will be permissible, provided this is part of local practice.
  Interventions: Procedure: Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy]
- CHRONOS A - Arm 2 (Intervention) (Experimental): Focal therapy alone (high intensity focused ultrasound [HIFU] or cryotherapy as per physician and centre choice). A second focal therapy session in-field, or a first focal therapy session to an out-of-field progressive or de novo lesion will be allowed as part of the focal therapy intervention.
  Interventions: Procedure: Focal therapy
- CHRONOS B - Arm 3 (Control) (Experimental): Focal therapy alone (high intensity focused ultrasound [HIFU] or cryotherapy as per physician and centre choice). A second treatment in-field, or a first focal ablation to an out-of-field progressive or de novo lesion will be allowed but will be regarded as failure events for the purpose of CHRONOS-B.
  Interventions: Procedure: Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy]
- CHRONOS B - Arm 4 (Intervention): (Experimental): Neoadjuvant finasteride 5mg once daily for a minimum of 12 weeks followed by focal therapy (as per CHRONOS B control arm).
  Interventions: Procedure: Focal therapy after Finasteride 5Mg tablets for 12 weeks
- CHRONOS B - Arm 5 (Intervention) (Experimental): Neoadjuvant bicalutamide 50mg once daily therapy for a minimum of 12 weeks followed by focal therapy (as per control arm).
  Interventions: Procedure: Focal therapy after Bicalutamide 50Mg tablets for 12 weeks

INTERVENTIONS:
Procedure: Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy] — Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy]
  Other Names: radiotherapy; prostatectomy; external beam radiotherapy; brachytherapy
  Arms: CHRONOS A - Arm 1 (Control); CHRONOS B - Arm 3 (Control)
Procedure: Focal therapy — Focal therapy (high intensity focused ultrasound or cryotherapy)
  Other Names: high intensity focused ultrasound; cryotherapy; HIFU
  Arms: CHRONOS A - Arm 2 (Intervention)
Procedure: Focal therapy after Finasteride 5Mg tablets for 12 weeks — finasteride 5mg tablets 12 weeks prior to focal therapy
  Other Names: Neoadjuvant
  Arms: CHRONOS B - Arm 4 (Intervention):
Procedure: Focal therapy after Bicalutamide 50Mg tablets for 12 weeks — Bicalutamide 50mg per day - 12 weeks prior to focal therapy
  Other Names: Neoadjuvant
  Arms: CHRONOS B - Arm 5 (Intervention)

SUMMARY:
Men diagnosed with significant cancer confined to the prostate currently undergo radical therapy directed to the whole prostate (radiotherapy or prostatectomy). These provide good cancer control but can cause significant side effects.

Focal Therapy involves targeting the cancer alone, whilst leaving healthy prostate gland alone. Case series have shown similar cancer control over 5 years with a much better side effect profile. However, there have been no randomised control trials (RCTs) comparing the success in cancer control and the quality of life in patients that undergo radical therapy vs those that undergo focal therapy. Further, there is a need to assess the use of additional therapies that may improve the cancer control outcomes following focal therapy. By having a trials platform with two RCTs (CHRONOS-A and CHRONOS-B) that reflect best patient and physician preferences/ equipoise, the investigators aim to answer these questions.

To improve acceptability, recruitment and compliance, the investigators have an embedded study aimed at reviewing clinician and patient perspectives and trial acceptability. CHRONOS-A will compare radical therapy to focal therapy, whilst CHRONOS-B will compare focal therapy alone to focal therapy with various therapies targeting the testosterone pathway that can shrink the cancer before it is treated. The investigators think this might improve outcomes further for men that definitely want focal therapy.

DETAILED DESCRIPTION:
AIM:

CHRONOS-A

Pilot: To determine if men will agree to participate in a randomised controlled trial that randomly assigns them to focal therapy alone or radical therapy (radiotherapy or prostatectomy).

Main: To determine if focal therapy alone is non-inferior when compared to radical therapy (radiotherapy or surgery) in terms of progression-free survival at 5 years in men with clinically significant non-metastatic cancer.

CHRONOS-B

Pilot: To determine if men expressing a preference for focal therapy will agree to participate in a multi-arm, multi-stage Randomised Controlled Trial that randomly assigns them to focal therapy alone or focal therapy in combination with neoadjuvant and/or adjuvant agents.

Main: To determine if focal therapy combined with neoadjuvant and/or adjuvant agents, compared to focal therapy alone, will improve failure-free survival at 5 years, in men with clinically significant non-metastatic cancer.

OBJECTIVES To deliver a trials framework that fits with existing patient and physician equipoise so that the investigators can answer the next generation of research questions to evaluate medium-term outcomes following minimally invasive focal therapy in the treatment of clinically significant, non-metastatic prostate cancer.

Embedded internal pilot objectives:

* Determine patient acceptance to randomisation.
* Conduct an embedded qualitative study of patient and clinician acceptance and experience of the linked randomised controlled trial CHRONOS design.
* Establish the feasibility of an economic evaluation alongside the main trial.
* Determine acceptability and completeness of resource use and utility measures.
* Identify the relevant NHS and non-NHS resource use to be collected alongside the main trial.
* Identify the relevant items to populate the Cost and Consequences framework.
* Perform preliminary analysis of pattern of missing data.

MAIN STUDY PRIMARY OBJECTIVES

CHRONOS-A:

To evaluate progression-free survival rates of focal therapy alone compared to radical therapy (radiotherapy or surgery) in the treatment of non-metastatic clinically significant prostate cancer. Progression-free survival is defined as time from randomisation to salvage whole-gland or systemic therapy, prostate cancer metastases or prostate cancer-specific mortality.

CHRONOS-B:

To evaluate Failure-Free-Survival rates of focal therapy alone compared to focal therapy combined with other therapies as a neoadjuvant strategy. Failure-Free-Survival is defined as time from randomisation to further focal therapy session or salvage whole-gland or systemic therapy or prostate cancer metastases or prostate cancer-specific mortality.

MAIN STUDY SECONDARY OBJECTIVES

Disease control:

Determine the histological, biochemical and oncological disease control for men undergoing radical therapy, focal therapy or focal therapy with neo/adjuvant treatments.

Adverse events and Functional Outcomes:

Determine the adverse events and functional outcomes after radical therapy, focal therapy or focal therapy with neo/adjuvant treatments

Health economics:

* Establish the NHS costs of the different interventions.
* Determine the Cost per QALYs (CUA), cost per PFS/FFS (CEA) and cost and consequences (CCA).
* Determine acceptability and completeness of resource use and utility measures.

Qualitative:

* Patient experience of consent and recruitment, including reasons for declining participation.
* Participants' motivation to accept randomisation to and compliance with an intervention, which may or may not include neoadjuvant and adjuvant treatments.
* Patients' understanding and experience of each trial arm.
* Patients' experience of toxicities, focusing on erectile dysfunction and urinary symptoms.
* Patients' attitudes to the predicted survival rate.
* Potential improvements to recruitment processes.
* Healthcare professionals' attitudes to intervention arms and trial design and whether this might impact on recruitment.

Imaging and Histology:

* Compare MRI outcomes with histology at time-points in which both are mandated.

Biobank and databank objectives:

* Evaluate cancer infiltrating immune cells and immune gene signatures following ablation.
* Build a biobank and databank of matched imaging, blood, serum, plasma and pre-digital rectal examination urine as well as FFPE biopsy samples.

DURATION :

Pilot: Recruitment 12 months. Minimum 3 months follow-up. Main study: Recruitment further 48 months. Total including follow-up = 96 months

SAMPLE SIZE :

Pilot Study - CHRONOS-A & B - 60 patients each over 12-months. Main study - CHRONOS-A - 1190 patients / CHRONOS-B - 1260 patients. PATIENT POPULATION: Men with non-metastatic prostate cancer who are suitable for focal therapy and radiotherapy.

PRIMARY ENDPOINTS (Main Stage) CHRONOS-A: Progression-Free survival (PFS) defined as biochemical failure (radical therapies only) or salvage therapy (local or systemic) or prostate cancer metastases or prostate cancer specific mortality.

CHRONOS-B: Failure-Free survival (FFS) defined as more than one focal therapy session or salvage therapy (local or systemic) or prostate cancer metastases or prostate cancer specific mortality.

SECONDARY ENDPOINTS (Main Stage)

Disease control:

* Rates of positive biopsy for any prostate cancer and significant cancer defined by a number of different thresholds on biopsy following focal therapy (treated and untreated side).
* Rates of second or third focal therapy sessions, in-field or out-of-field.
* Rates of radiotherapy as adjuvant or salvage therapy following surgery or focal therapy.
* Rates of prostatectomy as adjuvant or salvage therapy following radiotherapy or focal therapy.
* Rates of systemic therapy as adjuvant or salvage therapy following surgery, radiotherapy or focal therapy.
* Rates of prostate cancer-specific mortality.
* Rates of all-cause mortality.
* Long-term health outcomes of those participants consenting to longitudinal follow-up will be reported in subsequent studies pending further funding.

Adverse events and functional outcomes:

* Rates of cystoscopic interventions following treatment.
* Rates of implant insertion for treatment of incontinence and erectile dysfunction.
* Rates of medication and/or pump devices used for erectile dysfunction following treatment.
* Rates of endoscopic investigations of the lower bowel following treatment.
* Rates of pad-use and quantity per day for urinary incontinence following treatment.
* Rates of pad-use and quantity per day for faecal incontinence following treatment.
* Rates of adverse event rates and complications.
* Genito-urinary and rectal side-effects using patient-reported outcome measures using validated questionnaires including evaluation of return to baseline function for erectile and urinary function and various minimum decreases in PROMS scores.

Health economics:

* To establish the NHS costs of the different interventions.
* To determine the incremental cost per quality adjusted life year (QALYs)gained over the estimated lifetime of participants for focal therapy versus radical therapy.
* To determine the incremental cost per quality adjusted life year (QALYs) gained over the estimated lifetime of participants for focal therapy versus focal therapy with neoadjuvant and/or adjuvant strategies.

Qualitative:

* The impact on participants' overall health-related quality-of-life including adverse events and impact on genito-urinary and rectal functional status using validated patient reported outcome measures.
* Descriptive analyses of the questionnaire data, and use of questionnaire and qualitative interview datasets in a multi-methods analysis to look for overarching themes in barriers and facilitators to participation in CHRONOS-A and CHRONOS-B.

Imaging and Pathology

* Accuracy and variability of multi-parametric MRI (mpMRI) in detecting disease at baseline prior to focal therapy and absence or presence of recurrence of cancer based on histology outcomes on biopsy. Target definition for recurrence will be defined as significant prostate cancer as per inclusion criteria.

Translational, Biobank and Databank:

* Analysis on the localisation and nature of cancer-infiltrating immune cells and the immune-relevant gene expression within the cancer tissue.
* The creation of a biobank and databank of matched blood, serum, plasma and pre-digital rectal examination urine as well as imaging as well as FFPE biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

* PSA </=20ng/ml
* Patients must have undergone a diagnostic pre-biopsy MRI compliant with national uro-radiology consensus guidelines. Dynamic contrast enhancement using gadolinium is not required at diagnostic stage. However, contrast enhancement MRI will be required in those men who undergo focal therapy prior to focal therapy as a baseline for comparison during follow-up. In the absence of a compliant MRI (for clinical or other reasons), a transperineal template mapping biopsy using a 5-10 mm sampling frame will be required
* Histologically proven prostate adenocarcinoma
* Overall Gleason score of 7 (either 3+4=7 or 4+3=7) of any length or Gleason 3+3=6 provided >/=6mm cancer core length in any one core. Patients with Gleason 4+4=8 in some cores but where the overall Gleason score is 7 will be included.
* Bilateral histologically proven prostate cancer is permissible provided the following criteria are met:

  * The index lesion to be treated if focal therapy is used meets the above histological criteria.
  * The patient may have a PIRADS or Likert score 3, 4, 5 mpMRI lesion on the same hemi-gland (either right/left or anterior/posterior) as the histological index lesion
  * Secondary areas of Gleason 3+3=6 of </=5mm cancer outside of the treatment field can be monitored, if present, and patient undergoes focal therapy.
  * If a Likert or PIRADS score 3,4 or 5 mpMRI lesion is present in an area outside of the treatment field with a negative biopsy for cancer then pathology must be reviewed and confirm the presence of inflammation or atrophy if the patient is to undergo focal therapy*
* Radiological stage T2b/T3a will require central review regarding suitability for focal therapy.
* Index tumour volume, as seen on mpMRI if carried out, will be restricted to 50% of one lobe for either unilateral or bilateral ablation, patients with tumour volume >/=50% of one lobe will require central review prior to enrolment. Final decisions on suitability of focal therapy will lie with the trial central review in these cases.
* No restriction exists in CHRONOS-A on previous or current use of 5-alpha reductase inhibitors or anti-androgens or LHRH agonists or LHRH antagonists.
* Age at least 18 years of age
* Participants must be fit to undergo all procedures listed in the protocol as judged by clinical team

Exclusion Criteria:

* Previous or current LHRH agonist or LHRH antagonist or anti-androgen use in CHRONOS-B.
* Patients already established on a 5 alpha-reductase inhibitor (finasteride or dutasteride) who wish to go into CHRONOS-B will need to discontinue this for at least 6 months prior to randomisation. (NB: testosterone supplementation is permitted)
* Previous treatment for prostate cancer
* Life expectancy is likely to be less than 10 years
* Unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, Principal Investigator — Imperial College London
Locations (10):
- United Kingdom (10):
  - King's College Hospital NHS Foundation Trust, Brixton, London
  - West Middlesex Hospital, Isleworth, Middlesex
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, High Heaton, Newcastle Upon Tyne
  - Ashford & St Peter's Hospitals (ASPH) NHS Foundation Trust, Chertsey, Surrey
  - Hampshire Hospital NHS Foundation Trust, Basingstoke
  - Kingston Hospital NHS Foundation Trust, Kingston upon Thames
  - Imperial College Healthcare NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy D, Shah TT, Dudderidge T, McCracken S, Arya M, Dobbs C, Emberton M, Fiorentino F, Day E, Prevost AT, Staffurth J, Sydes M, Winkler M, Ahmed HU. Comparative Healthcare Research Outcomes of Novel Surgery in prostate cancer (IP4-CHRONOS): A prospective, multi-centre therapeutic phase II parallel Randomised Control Trial. Contemp Clin Trials. 2020 Jun;93:105999. doi: 10.1016/j.cct.2020.105999. Epub 2020 Apr 14. PMID 32302790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CHRONOS-A: At a conservative rate the two-arm RCT was expected to recruit 60 patients in the Pilot Stage in 6 centres over 12-months.
  CHRONOS-B: The three-arm MAMS RCT was expected to recruit 60 patients in the Pilot Stage in 6 centres over 12-months
Pre-assignment Details: CHRONOS A Arms have been combined as the Study aim was to determine if patients would agree to partake in an RCT that randomly assigns them to focal therapy alone or radical therapy
  CHRONOS B Arms have been combined as the Study aim was to determine if patients would agree to partake in an RCT that randomly assigns them to focal therapy alone or focal therapy in combination with neoadjuvant
Groups:
- CHRONOS A - Arm 1 (Control): CHRONOS-A was a two arm RCT.
  • Arm 1 (Control): Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy]). In patients undergoing radiotherapy, a maximum of 6-months neo-adjuvant hormonal therapy was allowed. In patients undergoing radical prostatectomy, cytoreduction a maximum of 6 months with medication was permissible, provided this was part of local practice.
- CHRONOS A - Arm 2 (Intervention): CHRONOS-B was a Multi-Arm Multi-Stage (MAMS) RCT.
  • Arm 2 (Intervention): Neoadjuvant finasteride 5mg once daily for a minimum of 12 weeks followed by focal therapy (as per control arm).
- CHRONOS B - Arm 4 (Intervention): Neoadjuvant finasteride 5mg once daily for a minimum of 12 weeks followed by focal therapy (as per CHRONOS B control arm).
  Focal therapy after Finasteride 5Mg tablets for 12 weeks: finasteride 5mg tablets 12 weeks prior to focal therapy
Period: Overall Study
Arm/Group | CHRONOS A - Arm 1 (Control) | CHRONOS A - Arm 2 (Intervention) | CHRONOS B - Arm 3 (Control) | CHRONOS B - Arm 4 (Intervention) | CHRONOS B - Arm 5 (Intervention)
Started | 18 | 18 | 22 | 21 | 21
Completed | 15 | 17 | 22 | 21 | 21
Not Completed | 3 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHRONOS A - Arm 1 (Control) | CHRONOS A - Arm 2 (Intervention) | CHRONOS B - Arm 3 (Control) | CHRONOS B - Arm 4 (Intervention): | CHRONOS B - Arm 5 (Intervention) | Total
Number analyzed (Participants) | 18 | 18 | 22 | 21 | 21 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.78 (7.64) | 69.28 (4.6) | 64.55 (7.0) | 66.52 (7.53) | 66.71 (6.80) | 66.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 18 | 18 | 22 | 21 | 21 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 13 | 14 | 17 | 15 | 67
  Mixed | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1 | 0 | 2
  Black | 0 | 0 | 1 | 1 | 1 | 3
  Other | 1 | 0 | 1 | 0 | 0 | 2
  Not Reported | 8 | 5 | 5 | 2 | 5 | 25
IMD Decile [Count of Participants; unit: Participants] — In order to get an area-based estimate of deprivation, the participants' postcodes were converted into an Index of Multiple Deprivation (IMD) score. The IMD is the established index of deprivation for England Wales which is based on detailed ward-level index of deprivation based on severe separate domains.The IMD is based on seven domains of deprivation: income, employment, health, education, crime, barriers to housing, and living environment. Decile 1 represents the most deprived 10% of areas, while decile 10 represents the least deprived 10%
  Participants
    Decile 1 | 0 | 0 | 0 | 2 | 0 | 2
    Decile 2 | 0 | 1 | 2 | 0 | 1 | 4
    Decile 3 | 1 | 1 | 1 | 0 | 1 | 4
    Decile 4 | 2 | 1 | 4 | 3 | 6 | 16
    Decile 5 | 2 | 2 | 4 | 3 | 4 | 15
    Decile 6 | 2 | 2 | 3 | 1 | 0 | 8
    Decile 7 | 2 | 4 | 1 | 2 | 3 | 12
    Decile 8 | 3 | 4 | 2 | 4 | 3 | 16
    Decile 9 | 3 | 1 | 4 | 2 | 2 | 12
    Decile 10 | 3 | 2 | 1 | 4 | 1 | 11
    Missing from eCRF | 0 | 0 | 0 | 0 | 0 | 0
Digital Rectal Examination [Count of Participants; unit: Participants]
  Yes | 6 | 9 | 7 | 7 | 8 | 37
  Normal Findings | 3 | 5 | 4 | 3 | 6 | 21
  Abnormal Findings | 3 | 4 | 3 | 4 | 2 | 16
  No | 12 | 8 | 15 | 14 | 13 | 62
  Missing from eCRF | 0 | 1 | 0 | 0 | 0 | 1
Current Medication [Count of Participants; unit: Participants]
  Yes | 11 | 12 | 13 | 15 | 12 | 63
  No | 5 | 3 | 9 | 6 | 9 | 32
  Missing from eCRF | 2 | 3 | 0 | 0 | 0 | 5
5 alpha-reductase inhibitor [Count of Participants; unit: Participants]
  Yes over (or equal to) 6 months ago | 0 | 0 | 0 | 1 | 0 | 1
  Yes within 6 months | 0 | 1 | 0 | 0 | 0 | 1
  No | 16 | 14 | 22 | 20 | 21 | 93
  Missing from eCRF | 2 | 3 | 0 | 0 | 0 | 5
Tumour Grade [Count of Participants; unit: Participants] — Tumour's Gleason Score has been used to grade the Tumours. The Gleason grading system refers to how abnormal the prostate cancer cells look and how likely the cancer is to advance and spread. A lower Gleason grade means that the cancer is slower growing and is less aggressive.
  Gleason 3+3 - low-grade cancer Gleason 3+4 - medium-grade cancer Gleason 4+3 - medium-grade cancer but higher than 3+4
  Participants
    Gleason 3+3 | 1 | 1 | 2 | 2 | 0 | 6
    Gleason 3+4 | 14 | 13 | 16 | 16 | 17 | 76
    Gleason 4+3 | 3 | 4 | 4 | 3 | 4 | 18
Local Stage [Count of Participants; unit: Participants] — TNM Staging system has been used for Local Stage. The T refers to the size of the tumour and how far it has spread into nearby tissue. T2 being smaller and T3a being larger. The letter 'a' referring to whether the tumour has spread across the prostate.
  Participants
    Clinical T2/Radiological stage <T3a | 18 | 18 | 20 | 19 | 18 | 93
    Radiological T3a | 0 | 0 | 2 | 2 | 3 | 7
Previous or current 5ARI use? [Count of Participants; unit: Participants] — 5ARI stands for 5α-Reductase inhibitors. This is also known as dihydrotestosterone blockers, they are a class of medications with antiandrogenic effects which are used primarily in the treatment of an enlarged prostate Population: Only CHRONOS A used 5ARI. This was an exclusion criteria for B
  Participants
    Yes: number analyzed (Participants) | 18 | 18 | 0 | 0 | 0 | 36
    Yes | 0 | 1 | 0 | 0 | 0 | 1
    No: number analyzed (Participants) | 18 | 18 | 0 | 0 | 0 | 36
    No | 18 | 17 | 0 | 0 | 0 | 35

OUTCOME MEASURES:

1. Primary Outcome: Pilot: Acceptance of Randomisation to Allocated Arm Within CHRONOS A & CHRONOS B
Description: To assess the acceptance of randomisation to the allocated arm within CHRONOS A & CHRONOS B separately using rates of compliance, and rates of withdrawal
Time Frame: 12 months
Population: The count of participants recruited and randomised per month per centre (CHRONOS-A and CHRONOS-B separately)
Measure: Count of Participants; unit: Participants
Groups:
- CHRONOS A - Arm 1 (Control): • Arm 1 (Control): Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy]). In patients undergoing radiotherapy, a maximum of 6-months neo-adjuvant hormonal therapy was allowed. In patients undergoing radical prostatectomy, cytoreduction a maximum of 6 months with medication was permissible, provided this was part of local practice.
- CHRONOS A - Arm 2 (Intervention): • Arm 2 (Intervention): Focal therapy alone (high intensity focused ultrasound [HIFU] or cryotherapy as per physician and centre choice). A second focal therapy session in-field, or a first focal therapy session to an out-of-field progressive or de novo lesion was allowed as part of the focal therapy intervention.
- CHRONOS B - Arm 3 (Control): • Arm 1 (Control): Focal therapy alone (high intensity focused ultrasound [HIFU] or cryotherapy as per physician and centre choice). A second treatment in-field, or a first focal ablation to an out-of-field progressive or de novo lesion was allowed but were regarded as failure events for the purpose of CHRONOS-B.
- CHRONOS B - Arm 4 (Intervention):: • Arm 2 (Intervention): Neoadjuvant finasteride 5mg once daily for a minimum of 12 weeks followed by focal therapy (as per control arm).
- CHRONOS B - Arm 5 (Intervention): Arm 3 (Intervention): Neoadjuvant bicalutamide 50mg once daily therapy for a minimum of 12 weeks followed by focal therapy (as per control arm).
Arm/Group | CHRONOS A - Arm 1 (Control) | CHRONOS A - Arm 2 (Intervention) | CHRONOS B - Arm 3 (Control) | CHRONOS B - Arm 4 (Intervention): | CHRONOS B - Arm 5 (Intervention)
Number analyzed (Participants) | 18 | 18 | 22 | 21 | 21
Participants
  Charing Cross Hospital | 4 | 0 | 11 | 10 | 11
  University Hospital Southampton NHS Foundation Trust | 11 | 8 | 8 | 9 | 5
  Sunderland Royal Hospital | 0 | 4 | 0 | 0 | 2
  Ashford & St Peter's Hospitals NHS Foundation Trust | 0 | 2 | 3 | 1 | 2
  Royal Marsden Hospital NHS Foundation Trust | 0 | 0 | 0 | 0 | 0
  Hampshire Hospital NHS Foundation Trust | 1 | 0 | 0 | 0 | 0
  Kingston Hospital NHS Foundation Trust | 0 | 0 | 0 | 1 | 0
  West Middlesex University Hospital | 2 | 3 | 0 | 0 | 1
  The Newcastle Upon Tyne Hospitals NHS Foundation Trust | 0 | 1 | 0 | 0 | 0
  King's College Hospital NHS Foundation Trust | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Pilot: Recruitment Rate to CHRONOS A & CHRONOS B and Their Corresponding 95% Confidence Intervals
Description: To estimate the recruitment rate to CHRONOS A & CHRONOS B and their corresponding 95% confidence intervals
  The recruitment rate is defined as number recruited (consented) over total number of patients approached.
Time Frame: 12 months
Population: Recruitment rates of CHRONOS-A and CHRONOS-B and their corresponding 95% confidence intervals
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CHRONOS B - Arm 4 (Intervention): * Arm 2 (Intervention): Neoadjuvant finasteride 5mg once daily for a minimum of 12 weeks followed by focal therapy (as per control arm).
Arm/Group | CHRONOS A - Arm 1 (Control) | CHRONOS A - Arm 2 (Intervention) | CHRONOS B - Arm 3 (Control) | CHRONOS B - Arm 4 (Intervention) | CHRONOS B - Arm 5 (Intervention)
Number analyzed (Participants) | 211 | 211 | 148 | 148 | 148
percentage of participants | 8.5 [5.1 to 13.1] | 8.5 [5.1 to 13.1] | 14.9 [9.6 to 21.6] | 14.2 [9 to 20.9] | 14.2 [9 to 20.9]

3. Primary Outcome: Pilot: Treatment Compliance to CHRONOS - A
Description: To determine the treatment compliance of patients to receiving the treatment they have been allocated to through randomisation within CHRONOS A only and corresponding 95% confidence interval.
  CHRONOS B results provided in a separate table
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHRONOS A - Arm 1 (Control) | CHRONOS A - Arm 2 (Intervention)
Number analyzed (Participants) | 18 | 18
percentage of participants | 72.2 [46.5 to 90.3] | 88.9 [65.3 to 98.6]

4. Primary Outcome: Pilot: Treatment Compliance (CHRONOS-B)
Description: To determine the treatment compliance of patients to receiving the treatment they have been allocated to through randomisation within CHRONOS B only and corresponding 95% confidence interval
  CHRONOS A results provided in a separate table
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHRONOS B - Arm 3 (Control) | CHRONOS B - Arm 4 (Intervention): | CHRONOS B - Arm 5 (Intervention)
Number analyzed (Participants) | 22 | 21 | 21
percentage of participants | 100 [84.6 to 100] | 100 [83.9 to 100] | 100 [83.9 to 100]

5. Primary Outcome: Drug Compliance to CHRONOS-B Only
Description: To determine patients drug compliance to allocated IMP treatment within randomisation of CHRONOS-B Arm 4 and Arm 5 only as CHRONOS -B Arm 3 is non-IMP.
  CHRONOS Arm A is not included as both arms are non-IMP
Time Frame: 12 months
Population: CHRONOS B- Arm 3 was not included in the analysis as it was the control and therefore non-IMP.
  CHRONOS A - Arm 1 & Arm 2 not included as they are non-IMP
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHRONOS B - Arm 4 (Intervention): | CHRONOS B - Arm 5 (Intervention)
Number analyzed (Participants) | 21 | 21
percentage of participants
  Returned empty blister packs | 33.3 [14.6 to 57] | 23.8 [8.2 to 47.2]
  Patients given the IMP | 100 [83.9 to 100] | 100 [83.9 to 100]

6. Primary Outcome: Pilot: Randomisation Rate to CHRONOS A & CHRONOS B and Their Corresponding 95% Confidence Intervals
Description: To estimate the randomisation rate to CHRONOS A & CHRONOS B and their corresponding 95% confidence intervals
  The Randomisation rate is defined as number of randomised patients over total number of patients recruited (consented)
Time Frame: 12 months
Population: Randomisation rates of CHRONOS-A and CHRONOS-B and their corresponding 95% confidence intervals
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHRONOS A - Arm 1 (Control) | CHRONOS A - Arm 2 (Intervention) | CHRONOS B - Arm 3 (Control) | CHRONOS B - Arm 4 (Intervention) | CHRONOS B - Arm 5 (Intervention)
Number analyzed (Participants) | 18 | 18 | 22 | 21 | 21
percentage of participants | 48.6 [31.9 to 65.6] | 48.6 [31.9 to 65.6] | 34.4 [22.9 to 47.3] | 32.8 [21.6 to 45.7] | 32.8 [21.6 to 45.7]

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Groups:
- CHRONOS A - Arm 2 (Intervention) Focal Therapy Alone: Focal therapy alone (high intensity focused ultrasound [HIFU] or cryotherapy as per physician and centre choice). A second focal therapy session in-field, or a first focal therapy session to an out-of-field progressive or de novo lesion will be allowed as part of the focal therapy intervention.
  Focal therapy: Focal therapy (high intensity focused ultrasound or cryotherapy)
- CHRONOS B - Arm 1 (Control) Focal Therapy Alone: Focal therapy alone (high intensity focused ultrasound [HIFU] or cryotherapy as per physician and centre choice). A second treatment in-field, or a first focal ablation to an out-of-field progressive or de novo lesion will be allowed but will be regarded as failure events for the purpose of CHRONOS-B.
  Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy]: Radical therapy (radiotherapy or prostatectomy [radiotherapy can be external beam or brachytherapy]
- CHRONOS B - Arm 2 (Intervention) Neoadjuvant Finasteride 5mg: Neoadjuvant finasteride 5mg once daily for a minimum of 12 weeks followed by focal therapy (as per CHRONOS B control arm).
  Focal therapy after Finasteride 5Mg tablets for 12 weeks: finasteride 5mg tablets 12 weeks prior to focal therapy
- CHRONOS B - Arm 3 (Intervention) Neoadjuvant Bicalutamide 50mg: Neoadjuvant bicalutamide 50mg once daily therapy for a minimum of 12 weeks followed by focal therapy (as per control arm).
  Focal therapy after Bicalutamide 50Mg tablets for 12 weeks: Bicalutamide 50mg per day - 12 weeks prior to focal therapy
Arm/Group | CHRONOS A - Arm 1 (Control) | CHRONOS A - Arm 2 (Intervention) Focal Therapy Alone | CHRONOS B - Arm 1 (Control) Focal Therapy Alone | CHRONOS B - Arm 2 (Intervention) Neoadjuvant Finasteride 5mg | CHRONOS B - Arm 3 (Intervention) Neoadjuvant Bicalutamide 50mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/22 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/18 | 3/22 | 0/21 | 3/21
Other Adverse Events (participants affected / at risk) | 2/18 | 6/18 | 10/22 | 12/21 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHRONOS A - Arm 1 (Control) (N=18) | CHRONOS A - Arm 2 (Intervention) Focal Therapy Alone (N=18) | CHRONOS B - Arm 1 (Control) Focal Therapy Alone (N=22) | CHRONOS B - Arm 2 (Intervention) Neoadjuvant Finasteride 5mg (N=21) | CHRONOS B - Arm 3 (Intervention) Neoadjuvant Bicalutamide 50mg (N=21)
Iatrogenic scrotal oedema (Primary) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraphimosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urosepsis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial Cellulitis and Related Condition (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visible haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Torsades de Pointes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection due to common bile duct stones (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Common bile duct stones (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aortic stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CHRONOS A - Arm 1 (Control) (N=18) | CHRONOS A - Arm 2 (Intervention) Focal Therapy Alone (N=18) | CHRONOS B - Arm 1 (Control) Focal Therapy Alone (N=22) | CHRONOS B - Arm 2 (Intervention) Neoadjuvant Finasteride 5mg (N=21) | CHRONOS B - Arm 3 (Intervention) Neoadjuvant Bicalutamide 50mg (N=21)
Abdominal pain (Gastrointestinal disorders) | 1/14 (1) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Allergic reaction to Penicillin (Immune system disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Aortic stenosis (Cardiac disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Bacterial Cellulitis and Related Conditions (Infections and infestations) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Blood from urethral meatus when straining (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Campylobacter (Infections and infestations) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Chest infection (Infections and infestations) | 0/14 (0) | 1/16 (1) | 0/21 (0) | 0 (0) | 0 (0)
Complications of urinary catheter (Infections and infestations) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
COVID (Immune system disorders) | 0/14 (0) | 1/16 (1) | 0/21 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Dry ongoing cough, Chest xray clear (General disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Dry Orgasm (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Ejaculatory dysfunction (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Elective (planned) parathyroidectomy (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Epididymo-orchitis (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Erectile Dysfunction (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 6/21 (6) | 3 (3) | 6 (6)
Failed removal of common bile duct stones (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 2 (2) | 0 (0)
Haemtospermia (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/14 (0) | 1/16 (1) | 0/21 (0) | 0 (0) | 0 (0)
Iatrogenic Scrotal Oedema (Renal and urinary disorders) | 0/14 (0) | 1/16 (1) | 0/21 (0) | 0 (0) | 0 (0)
Infection following tooth extraction (Infections and infestations) | 0/14 (0) | 1/16 (1) | 0/21 (0) | 0 (0) | 0 (0)
Knee Replacement (General disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Low urinary flow rate (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 3/21 (3) | 1 (1) | 0 (0)
Nocturia (General disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Painful nipples (General disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Painless swelling and mild bruising of scrotal and penile skin (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
pancytopenia (Blood and lymphatic system disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Paraphimosis (Renal and urinary disorders) | 1/14 (1) | 0/16 (0) | 0/21 (0) | 0 (0) | 0 (0)
bladder malignancy (Renal and urinary disorders) | 1/14 (1) | 0/16 (0) | 0/21 (0) | 0 (0) | 0 (0)
patient required TURP after urosepsis and retention (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Penile numbness (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Penile tip pain (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Pleuritic Chest Pain - Bilateral pulmonary emboli on CT imaging (Cardiac disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Post HIFU Prostate Inflammation (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Post traumatic stress disorder (Psychiatric disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Prostatitis (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Reaction to Ciprofloxacin (Nausea and Vomiting) (General disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Rectal fissure (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Removal of stones from common bile duct (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Severe LUTS (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Short term memory loss (Psychiatric disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
stroke (Cardiac disorders) | 0/14 (0) | 1/16 (1) | 0/21 (0) | 0 (0) | 0 (0)
Suspected common bile duct stone/pancreatitis,serum amylase raised (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Sweaty testicles (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Swollen testicles (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
Torsades de Pointes (Cardiac disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Urgency of micturition (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1/14 (1) | 0/16 (0) | 1/21 (1) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 0/14 (0) | 1/16 (1) | 2/21 (2) | 1 (1) | 9 (9)
Urine leaking around catheter - ?catheter blocked, requires flushing. (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)
UTI, epididymo-orchitis (Infections and infestations) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 1 (1) | 0 (0)
Visible haematuria (Renal and urinary disorders) | 0/14 (0) | 0/16 (0) | 0/21 (0) | 0 (0) | 2 (2)
Worsening night sweats (General disorders) | 0/14 (0) | 0/16 (0) | 1/21 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04049747/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04049747/SAP_001.pdf